CLINICAL TRIAL: NCT07157410
Title: Two-year Clinical Evaluation of Different Indirect Tooth-colored Onlay Restorations Placed in Posterior Teeth With Cervical Margin Relocation and Laboratory Investigation of Marginal Adaptation
Brief Title: Clinical Evaluation of Indirect Tooth-Colored Onlays With Cervical Margin Relocation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A0502025CD
Record Dates: First submitted 2025-05-05; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-03

CONDITIONS: Indirect Tooth-colored Onlay Restorations in Posterior Teeth; Clinical Performance of Cervical-margin-relocated Onlay Restorations
Keywords: cervical margin relocation; marginal adaptation; Indirect onlay restorations; Lithium-disilicate; CAD/CAM composite
MeSH Terms: interventions — IPS e.max Press

STUDY DESIGN:
Intervention Model Description: Split-mouth randomized allocation at the tooth level (each participant receives three onlays, one per material).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Machinable lithium-disilicate ceramic onlay (IPS e.max CAD) (Experimental): Each participant contributes one randomized molar restored with a machinable lithium-disilicate onlay (IPS e.max CAD). Adhesive luting is performed under rubber-dam isolation using the standardized protocol.
  Interventions: Other: Machinable lithium-disilicate ceramic onlay (IPS e.max CAD)
- Pressed lithium-disilicate ceramic onlay (IPS e.max Press) (Experimental): Each participant contributes one randomized molar restored with a pressed lithium-disilicate onlay (IPS e.max Press). Adhesive luting is performed under rubber-dam isolation using the standardized protocol.
  Interventions: Other: Pressed lithium-disilicate ceramic onlay (IPS e.max Press)
- Machinable composite onlay (BRILLIANT Crios) (Experimental): Each participant contributes one randomized molar restored with a machinable composite onlay (BRILLIANT Crios). Adhesive luting is performed under rubber-dam isolation using the standardized protocol.
  Interventions: Other: Machinable composite onlay (BRILLIANT Crios)

INTERVENTIONS:
Other: Machinable lithium-disilicate ceramic onlay (IPS e.max CAD) — Single indirect onlay restoration milled from an IPS e.max CAD block and crystallized according to the manufacturer's Instructions for Use, then adhesively luted on a randomized molar under.
  Arms: Machinable lithium-disilicate ceramic onlay (IPS e.max CAD)
Other: Pressed lithium-disilicate ceramic onlay (IPS e.max Press) — Single indirect onlay restoration heat-pressed from an IPS e.max Press ingot and then adhesively luted on a randomized molar under rubber-dam isolation.
  Arms: Pressed lithium-disilicate ceramic onlay (IPS e.max Press)
Other: Machinable composite onlay (BRILLIANT Crios) — Single indirect onlay restoration milled from a BRILLIANT Crios block and then adhesively luted on a randomized molar under rubber-dam isolation.
  Arms: Machinable composite onlay (BRILLIANT Crios)

SUMMARY:
This study will evaluate the performance of three different tooth-colored onlay materials in adult patients' posterior teeth. First, investigators will use a bulk-fill composite resin to raise the cavity margin above the gum line and below the contact point. Then each patient will receive three onlays made from different materials. Investigators will follow patients at 2 weeks, 6 months, 18 months, and 24 months to assess how well the onlays fit, function, and whether restorations cause sensitivity or new decay. The results will help dentists choose the most durable onlay restorations for deep-margin elevation cases.

ELIGIBILITY:
Inclusion Criteria:

1. Molar tooth with proximal subgingival carious lesion of ICDAS 4 or 5, causing weakening of one or more cusps.
2. Normal alignment with the adjacent and opposing teeth.
3. Acceptance of the follow-up period and recall visits for 2 years.

Exclusion Criteria:

1. Distance between the gingival margin and the crestal bone < 2 mm.
2. The tooth would require direct pulp capping.
3. Poor oral hygiene (or not completing the oral hygiene phase).
4. Chronic periodontitis.
5. Pulpitis or non-vital tooth.
6. Orthodontic treatment.
7. Parafunctional habits.
8. Systemic disease.
9. Pregnancy.
10. Teeth act as abutment for fixed or removable prosthesis.
11. Occlusion of fewer than 20 teeth

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
FDI criteria score-functional (F1 Fracture/Retention; F2 Marginal Adaptation), biological (B1-B3), and miscellaneous (M2) domains. | Post-cementation baseline (2 weeks), 6, 12, 18, and 24 months
  Each onlay will be scored per the Revised 2023 World Dental Federation (FDI) criteria across the specified domains (F1, F2, B1, B2, B3, M2). Outcomes will be summarized as (a) mean (SD) score for each domain, and (b) proportion of restorations rated 1-3 (clinically acceptable) vs 4-5 for each domain. Lower scores indicate better clinical performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt